CLINICAL TRIAL: NCT02715531
Title: An Open-Label, Multicenter Phase Ib Study of The Safety and Efficacy of Atezolizumab (Anti-PD-L1 Antibody) Administered in Combination With Bevacizumab and/or Other Treatments in Patients With Solid Tumors
Brief Title: A Study of the Safety and Efficacy of Atezolizumab Administered in Combination With Bevacizumab and/or Other Treatments in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO30140
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Fluorouracil; atezolizumab; Bevacizumab; Gemcitabine; Leucovorin; 130-nm albumin-bound paclitaxel; Oxaliplatin; Capecitabine; Cisplatin

ARMS (5):
- Arm A (Hepatocellular Carcinoma [HCC], All subtypes) (Experimental): Participants with advanced or metastatic and/or unresectable HCC who have received no prior treatment are non-randomized and will receive atezolizumab and bevacizumab, every 3 weeks (q3w), each cycle of 21 days, as long as participants are experiencing clinical benefit in the opinion of the investigator.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Arm B (Gastric Cancer) (Experimental): Participants with previously untreated human epidermal growth factor receptor 2 (HER2)-negative adenocarcinoma of the stomach or gastroesophageal junction (GEJ) are non-randomized and will receive atezolizumab, bevacizumab, and FOLFOX (oxaliplatin, leucovorin, and 5-fluorouracil [FU]), every 2 weeks (q2w), each cycle of 28 days, as long as participants are experiencing clinical benefit in the opinion of the investigator. Oxaliplatin will be administered for up to 8 cycles. After 6 months, at discretion of investigator, capecitabine may be administered as maintenance therapy without oxaliplatin instead of infusional 5-FU and leucovorin, and biologic therapy may be given every 3 weeks (q3w). In the event that a patient experiences unacceptable toxicity after replacement of infusional 5-FU and leucovorin with capecitabine, the patient may be allowed to switch back to 5-FU and leucovorin following investigator discussion with the Medical Monitor.
  Interventions: Drug: 5-FU; Drug: Atezolizumab; Drug: Bevacizumab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Capecitabine
- Arm C (Metastatic Pancreatic Cancer) (Experimental): Participants with previously untreated metastatic pancreatic cancer are non-randomized and will receive atezolizumab q2w starting on Day 1, Cycle 1 (each cycle of 28 days). Administration of nab-paclitaxel followed by gemcitabine will occur on Days 1, 8, and 15 of each cycle (3-weeks-on/1-week-off schedule). Treatment consisting of atezolizumab with gemcitabine and nab-paclitaxel may be continued as long as participants are experiencing clinical benefit in the opinion of the investigator.
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Nab-Paclitaxel
- Arm E (Randomized Metastatic Esophageal Cancer) (Experimental): Participants with squamous metastatic esophageal cancer (mEC) will be randomized (1:1) into Group E1 and Group E2. All participants with metastatic adenocarcinoma of esophageal carcinoma or GEJ Siewert Classification Type I will be enrolled into Group E3. In Groups E1 and E3, participants will receive atezolizumab and FOLFOX, q2w, each cycle of 28 days, as long as participants are experiencing clinical benefit in opinion of the investigator. Oxaliplatin will be administered for up to 8 cycles. In Group E2, participants will receive atezolizumab followed by cisplatin and 5-FU q3w. Cisplatin will be administered for up to 6 cycles. Treatment with atezolizumab in combination with 5-FU may be continued as long as participants experience clinical benefit in opinion of the investigator.
  Interventions: Drug: 5-FU; Drug: Atezolizumab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Cisplatin
- Arm F (Randomized HCC) (Experimental): Participants with advanced or metastatic and/or unresectable HCC who have received no prior systemic treatment will be randomized (1:1) into Group F1 and Group F2. Participants will receive atezolizumab alone (Group F2) or combined with bevacizumab (Group F1) on a q3w schedule, with dosing on Day 1 of each 21 day Cycle. Treatment with atezolizumab with or without bevacizumab may be continued as long as participants are experiencing clinical benefit in the opinion of the investigator. Participants who are randomly assigned to Group F2 (atezolizumab monotherapy) and experience investigator-assessed unequivocal radiographic progression as per RECIST v1.1 will also be given the option to cross over to atezolizumab and bevacizumab combination therapy, provided they meet the criteria for crossover and Medical Monitor approval is obtained.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: 5-FU — 5-FU (400 mg/m^2) will be administered as an IV bolus, followed by 2400 mg/m^2 by continuous IV infusion over 46 (± 1) hours, q2w.
  Arms: Arm B (Gastric Cancer); Arm E (Randomized Metastatic Esophageal Cancer)
Drug: Atezolizumab — Participants will receive atezolizumab in a flat dose of 1200 mg q3w (Arm A, Group E2, and Arm F) or 840 mg q2w (Arm B, Arm C, and Groups E1 and E3).
  Other Names: Tecentriq; RO5541267
Drug: Bevacizumab — Participants will receive bevacizumab at 15 mg/kg q3w (Arm A and Group F1) or 10 mg/kg q2w (Arm B).
  Arms: Arm A (Hepatocellular Carcinoma [HCC], All subtypes); Arm B (Gastric Cancer); Arm F (Randomized HCC)
Drug: Gemcitabine — Gemcitabine will be administered according to the local prescribing information. The starting dose-level of gemcitabine (1000 mg/m^2) will be administered intravenously over 35 (± 5) minutes on Days 1, 8, and 15 of each 28-day cycle (3-weeks-on/1-week-off schedule).
  Arms: Arm C (Metastatic Pancreatic Cancer)
Drug: Leucovorin — Leucovorin 200 mg/m^2 L-isomer form or 400 mg/m^2 D,L-racemic form will be administered IV over 120 (± 15) minutes, q2w.
  Arms: Arm B (Gastric Cancer); Arm E (Randomized Metastatic Esophageal Cancer)
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered according to the local prescribing information. The starting dose-level of nab-paclitaxel (125 mg/m^2) will be administered intravenously over 35 (± 5) minutes on Days 1, 8, and 15 of each 28-day cycle (3-weeks-on/1-week-off schedule).
  Arms: Arm C (Metastatic Pancreatic Cancer)
Drug: Oxaliplatin — Oxaliplatin 85 mg/m^2 will be administered IV over 120 (± 5) minutes q2w.
  Arms: Arm B (Gastric Cancer); Arm E (Randomized Metastatic Esophageal Cancer)
Drug: Capecitabine — Capecitabine may be administered after 6 months at the discretion of the investigator (range of 650-1000 mg/m^2) twice daily on Days 1-4 of a 21-day cycle.
  Arms: Arm B (Gastric Cancer)
Drug: Cisplatin — Cisplatin will be administered as 80 mg/m^2 IV over 120 minutes q3w (Group E2).
  Arms: Arm E (Randomized Metastatic Esophageal Cancer)

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of atezolizumab in combination with bevacizumab, bevacizumab + oxaliplatin, leucovorin and 5-fluorouracil (5-FU) (FOLFOX), vanucizumab, nab-paclitaxel + gemcitabine, FOLFOX, or 5-FU + cisplatin, in participants with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion criteria

* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function
* Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade less than or equal to (</=) 1 prior to study entry, with the exception of alopecia
* Ready to use reliable contraceptive procedures

Inclusion Criteria Specific to HCC (Arm A and Arm F):

* Participants with advanced or metastatic and/or unresectable HCC
* The participant has disease that is not amenable to a curative approach
* No prior line of systemic therapy (includes participants who are sorafenib-naïve)
* Willing to undergo fresh liver biopsy if provided archival tissue was taken greater than (>) 6 months from Cycle 1 Day 1
* Child-Pugh Score of up to B7
* Serum bilirubin </= 3 times upper limit of normal (x ULN)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) </= 2 x ULN
* Albumin >2.8 grams per deciliter (g/dL)
* Documented virology status of hepatitis, as confirmed by screening hepatitis B surface antigen (HBsAg), antibody to hepatitis B core antigen (anti-HBc), and/or anti-hepatitis C virus (anti-HCV)
* Antiviral therapy per local standard-of-care if active hepatitis B virus (HBV)

Inclusion Criteria Specific to Arm A (Patients must also meet all of the following specific inclusion criteria to be eligible for enrollment in Arm A:)

* Child-Pugh score of up to B7
* Willing to undergo biopsy if archival tissue is not available or if archival tissue was taken >6 months from Cycle 1, Day 1
* Anti-viral therapy per local standard-of-care if active hepatitis B virus (HBV).

Inclusion Criteria Specific to Arm F (Patients must also meet all of the following specific inclusion criteria to be eligible for enrollment in Arm F:)

* LIfe expectancy >=3 months, as determined by the investigator
* Child-Pugh score A
* Platelet count ≥ 75x109/L (75,000/uL) without transfusion
* Availability at the site of tumor specimens in paraffin blocks (preferred) or 16 unstained slides, with an associated pathology report, prior to study entry
* Anti-viral therapy per local standard-of-care if active hepatitis B virus (HBV).

Inclusion Criteria Specific to Gastric Cancer (Arm B) (Patients must also meet all of the following specific inclusion criteria to be eligible for enrollment in Arm B:)

* Histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the stomach or GEJ in participants who have not received prior systemic therapy for metastatic disease
* Absence of HER2 expression documented as in situ hybridization (ISH) negative on previously collected and assessed tumor tissue upon initial diagnosis of disease

Inclusion criteria specific to metastatic pancreatic cancer (Arm C) (Patients must also meet all of the following specific inclusion criteria to be eligible for enrollment in Arm C:)

* Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas
* No previous radiotherapy, surgery, chemotherapy, or investigational therapy for the treatment of metastatic disease

Inclusion Criteria Specific to mEC (Arm E) (Patients must also meet all of the following specific inclusion criteria to be eligible for enrollment in Arm E:)

* Histologically or cytologically confirmed locally mEC or metastatic adenocarcinoma of the GEJ Siewert Classification Type I in participants who have not received prior systemic therapy for primary and metastatic disease or chemoradiation therapy for primary disease
* Absence of HER2 expression documented as ISH-negative on previously collected and assessed tumor tissue upon initial diagnosis of disease
* Willing to undergo biopsy if archival tissue is not available or if archival tissue was taken >6 months from Cycle 1 Day 1

Exclusion Criteria:

General Exclusion Criteria

* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease (exception for participants in Arm A and Arm F)
* Known primary central nervous system (CNS) malignancy or untreated or active CNS metastases
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or other recombinant human antibodies
* Positive test for Human Immunodeficiency Virus (HIV)
* Active hepatitis B (chronic or acute), or hepatitis C (exception for participants in Arm A and Arm F)
* Active tuberculosis
* Severe infections within 4 weeks prior to Day 1
* Signs or symptoms of significant infection within 2 weeks prior to Day 1
* Received oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1
* Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to Day 1, unstable arrhythmias, or unstable angina
* History of stroke, reversible ischemic neurological defect or transient ischemic attack within 6 months prior to Day 1
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's and/or Medical Monitor's judgment, precludes the participants safe participation in and completion of the study
* Malignancies other than pancreatic carcinoma within 2 years prior to study start, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent)

Exclusion Criteria Related to Medications

* Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA4), anti-programmed death-1 (anti-PD-1), or anti-programmed death ligand-1 (anti-PD-L1) therapeutic antibody
* Treatment with systemic immunostimulatory agents within 6 weeks or five half-lives of the drug, whichever is longer, prior to screening
* Treatment with systemic corticosteroids or other immunosuppressive medications within 2 weeks prior to Cycle 1, Day 1
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Participants with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Known allergies to oxaliplatin (or other platinum agents), leucovorin, 5-FU, nab-paclitaxel (or other taxanes) or gemcitabine

Exclusion Criteria Specific to Bevacizumab-Containign Arms (Arms A, B, and F) (Patients who meet any of the following criteria will be excluded from enrollment into bevacizumab-containing Arms A, B, and F:)

* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to the first dose of bevacizumab or vanucizumab
* History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to Day 1
* History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction within 6 months prior to Day 1 of Cycle 1
* Clinical signs or symptoms of GI obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
* Proteinuria, as demonstrated by urine dipstick or > 1.0 g of protein in a 24-hour urine collection
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses of large volume. HCC participants (Arm A and F) with vascular invasion of the portal or hepatic veins may be enrolled
* History of intra-abdominal inflammatory process within 6 months prior to Day 1 of Cycle 1
* Radiotherapy within 28 days and abdominal/pelvic radiotherapy within 60 days prior to Day 1 of Cycle 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1
* Chronic daily treatment with a nonsteroidal anti-inflammatory drug (NSAID)

Exclusions specific to Arms A and F (HCC) (Patients who meet any of the following specific exclusion criteria will be excluded from enrollment in Arms A and F:)

* Participants with untreated or incompletely treated varices with bleeding or high-risk for bleeding
* Treatment with any HCV anti-viral therapy within 4 weeks prior to Cycle 1 Day 1
* Moderate or severe ascites
* Hepatic encephalopathy

Exclusion Criteria Specific to Arm B (Gastric Cancer) (Patients who meet any of the following specific exclusion criteria will be excluded from enrollment in Arm B:)

* HER2 expression as defined by ISH positive and/or 3+ by immunohistochemistry (IHC)
* Prior treatment with an oxaliplatin-containing regimen
* Previous antiangiogenic therapy
* Ongoing treatment for epilepsy

Exclusion Criteria Specific to Arm C (Metastatic Pancreatic Cancer) (Patients who meet any of the following specific exclusion criteria will be excluded from enrollment in Arm C:)

* Patients with only locally advanced disease
* Presence of islet cell neoplasms

Exclusions Specific to Arm E (Metastatic Esophageal Cancer) (Patients who meet any of the following specific exclusion criteria will be excluded from enrollment in Arm E:)

* HER2 expression as defined by ISH positive and/or 3+ by immunohistochemistry
* Prior chemotherapy treatment, including radio-sensitization in pre- and post-operative settings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With At Least One Adverse Event, with Severity Determined According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | From screening to up to 90 days after the last dose of study drug (up to approximately 55 months)
Percentage of Participants with Objective Response as Determined By The Independent Review Facility (IRF) According To Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (Arm A) | From screening to end of study (approximately 55 months)
Progression-Free Survival (PFS) as determined by the Independent Review Facility (IRF) according to RECIST v 1.1 (Arm F) | From randomization to the first occurrence of disease progression or death from any cause (whichever occurs first)

SECONDARY OUTCOMES:
Serum Concentrations of Atezolizumab (All Arms) | Predose (0 hour[h]), 30 minutes(min) postdose on Day 1 of Cycles(Cy) 1 and 3; Predose(0h) on Day 1 of Cy 2,4,8 and every 8 Cy until treatment discontinuation (up to 55 months); 120 days after last dose (Cy length=21-28 days; up to 55 months)
Serum Concentrations of Bevacizumab (Arm A, Arm B and Group F1) | Predose (0 h) and 30 min postdose (infusion length=30-90 min) on Day 1 of Cy 1 and 3; at treatment discontinuation (up to 55 months); at 120 days after last dose (Cy length=21-28 days; up to 55 months)
Plasma Concentration of Oxaliplatin (Arm B and Group E1) | Predose (0 h) and 5-10 min before the end of infusion (infusion length=120 min) on Day 1 of Cycles 1 and 3 (Cycle length=21-28 days; up to approximately 3 months)
Plasma Concentration of 5-FU (Arm B and Arm E) | Predose (0 h), immediately following bolus administration and 2 hours post-bolus dose on Day 1 of Cycles 1 and 3 (Cycle length=21-28 days; up to approximately 3 months)
Plasma Concentration of Cisplatin (Group E2) | Predose (0 h) and 5-10 minutes before the end of infusion (infusion length=120 min) on Day 1 of Cycles 1 and 3 (Cycle length=21 days; up to approximately 3 months)
Plasma Concentration of nab-Paclitaxel (Arm C) | Predose (0 h), 5-10 minutes before the end of infusion and 1 hour after the end of the infusion (infusion length=35 min) on Day 1 of Cycles 1 and 3 (Cycle length=28 days; up to approximately 3 months)
Plasma Concentration of Gemcitabine (Arm C) | Predose (0 h), 5-10 minutes before the end of infusion and 1 hour after the end of the infusion (infusion length=35 min) on Day 1 of Cycles 1 and 3 (Cycle length=28 days) (up to approximately 3 months)
Percentage of Participants with Objective Response as Determined by the IRF according to RECIST v 1.1 (Arm F) | Baseline, every 8 weeks (± 1 week) for the first 12 months following Cycle 1 Day 1, and every 12 weeks (± 1 week) thereafter up to study completion (Cycle length=21-28 days; up to approximately 55 months)
Percentage of Participants with Objective Response as Determined By The Investigator According To RECIST v 1.1 (Arm A and Arm F) | Baseline, every 8 weeks (± 1 week) for the first 12 months following Cycle 1 Day 1, and every 12 weeks (± 1 week) thereafter up to study completion (Cycle length=21-28 days; up to approximately 55 months)
Percentage of Participants with Objective Response as Determined by the IRF according to HCC-Specific Modified RECIST (mRECIST) (Arm A and Arm F) | Baseline, every 8 weeks (± 1 week) for the first 12 months following Cycle 1 Day 1, and every 12 weeks (± 1 week) thereafter up to study completion (Cycle length=21-28 days; up to approximately 55 months)
Duration of Objective Response as Determined by the IRF according to RECIST v1.1 (Arm A and Arm F) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever comes first (up to approximately 55 months)
Duration of Objective Response as Determined by The Investigator According to RECIST v 1.1 (Arm A and Arm F) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever comes first (up to approximately 55 months)
Duration of Objective Response as Determined by the IRF According to HCC-Specific mRECIST (Arm A and Arm F) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever comes first (up to approximately 55 months)
PFS Duration as Determined by The IRF According to RECIST v1.1 (Arm A) | From the first dose of study treatment to the first occurrence of disease progression or death from any cause, whichever comes first (up to approximately 55 months)
PFS Duration as Determined by the Investigator According To RECIST v 1.1 (Arm A and Arm F) | From the first dose of study treatment (Arm A) or randomization (Arm F) to the first occurrence of disease progression or death from any cause, whichever comes first (up to approximately 55 months)
PFS Duration as Determined by the IRF Acording to HCC-Specific mRECIST (Arm A and Arm F) | From the first dose of study treatment (Arm A) or randomization (Arm F) to the first occurrence of disease progression or death from any cause, whichever comes first (up to approximately 55 months)
Overall Survival (OS) Duration (Arm A and Arm F) | Baseline up to study completion or death, whichever occurs first (up to approximately 55 months)
Time to Radiological Progression (TTRP) as Determined by the IRF According to RECIST v1.1 (Arm A and Arm F) | From the first dose of study treatment (Arm A) or randomization (Arm F) to the first occurrence of radiographic disease progression (up to approximately 55 months)
TTRP as Determined by The Investigator According to RECIST (Arm A and Arm F) | From the first dose of study treatment (Arm A) or randomization (Arm F) to the first occurrence of radiographic disease progression (up to approximately 55 months)
TTRP as Determined by The IRF According to HCC-Specific mRECIST (Arm A and Arm F) | From the first dose of study treatment (Arm A) or randomization (Arm F) to the first occurrence of radiographic disease progression (up to approximately 55 months)
Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) | Predose (0 h) on Day 1 of Cycles 1, 2, 3, 4, 8 and every 8 cycles until treatment discontinuation (up to 55 months); at 120 days after last dose (Cycle length =21-28 days; up to 55 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (12):
  - Stanford Cancer Institute; Hematology, Palo Alto, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
- The 81st Hospital of P.L.A., Nanjing, China
- Japan (4):
  - National Cancer Center Hospital East, Chiba
  - Yokohama City University Medical Center, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - The Cancer Institute Hospital of JFCR, Tokyo
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (5):
  - China Medical University Hospital, North Dist.
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - LINKOU; Dept of Cardiology, Taoyuan

REFERENCES:
- [Derived] Lee MS, Ryoo BY, Hsu CH, Numata K, Stein S, Verret W, Hack SP, Spahn J, Liu B, Abdullah H, Wang Y, He AR, Lee KH; GO30140 investigators. Atezolizumab with or without bevacizumab in unresectable hepatocellular carcinoma (GO30140): an open-label, multicentre, phase 1b study. Lancet Oncol. 2020 Jun;21(6):808-820. doi: 10.1016/S1470-2045(20)30156-X. PMID 32502443